CLINICAL TRIAL: NCT05802576
Title: Study of Interference Between Oral Anticoagulants and Heparin During Ablation of Atrial Fibrillation (AF) or Left Atrial Tachycardia (GAD) by Catheter
Acronym: FACADO
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP201314
Record Dates: First submitted 2023-03-27; First posted 2023-04-06 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Atrial Fibrillation; Atrial Tachycardia
Keywords: Atrial Fibrillation; Left Atrial Tachycardia; direct oral anticoagulants; unfractionated heparin
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Sample type : plasma. Quantity: 500. Plasma samples from blood samples will be frozen and will therefore be the subject of a biological collection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Vitamin K: The vitamin K oral anticoagulant will be used on 25 patients.
- Apixaban: The apixaban oral anticoagulant will be used on 25 patients.
- Rivaroxaban: The rivaroxaban oral anticoagulant will be used on 25 patients.
- Dabigatran: The dabigatran oral anticoagulant will be used on 25 patients.

SUMMARY:
Catheter ablation of atrial fibrillation (AF) or left atrial tachycardia (GAD) is usually performed in patients treated with vitamin K antagonists (VKAs) or direct oral anticoagulants (DOACs) that are increasingly used. In some cases, patients need to have an unfractionated heparin relay (UFH) for the procedure. There are no recommendations for adjusting UFH doses during an AOD/UFH relay. DOACs interfere with the biological assay of UFH which poses a problem of adaptation of UFH doses in pre- and intra-procedure. The aim of the study is to evaluate the interference of residual DOAC on the measurement of anticoagulant activity of UFH in pre- and intra-procedure of AF ablation or GAD.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is the most common heart rhythm disorder worldwide and is a major public health problem due to its increased morbidity and overall mortality, particularly related to stroke and heart failure. Catheter ablation is the most effective method for maintaining sinus rhythm and is currently recommended after failure of antiarrhythmic therapy in patients with symptomatic AF.

Spontaneous Atrial Left Tachycardia (ALT) is rarer, but is a common consequence after an initial procedure of persistent AF removal. The removal of AF, like that of ALT, is performed in the left atrium and is therefore associated with a major thromboembolic risk. The anticoagulation problems are the same for all ablations in the left atrium. Catheter ablation in the left atrium is usually performed in patients treated with vitamin K antagonists (VKAs) or direct oral anticoagulants (DOACs) that are increasingly used. In France, these are rivaroxaban and apixaban which are direct and selective inhibitors of factor Xa and dabigatran which directly and selectively inhibits free or clot-bound thrombin (factor IIa). DOACs are easier to use than VKAs and do not require regular biological monitoring either at initiation or in the follow-up of treatment. Based on current evidence from the AF literature, DOACs are comparable to VKAs with a lower risk of major bleeding.

Catheter ablation of AF or ALT exposes the patient to a hemorrhagic risk (hemopericardium for example) and especially thrombotic in intra-procedure ranging from 0.9 to 5%. Different mechanisms could be involved in this per-procedural prothrombotic situation: (1) activation of the contact phase by the ablation equipment, (2) lesion of the left atrial endothelium and release of pro-thrombotic cytokines from damaged cells, inflammatory reaction induced by the passage of transseptal sheaths (3) modification of blood flow after conversion to sinus rhythm. These different phenomena lead to the activation of coagulation. Conversely, excessive per-procedural anticoagulation exposes to a risk of bleeding. The management of patients under VKA is well codified and validated. In contrast, DOA treatment management is based solely on extrapolation of VKA data. Only a few observational studies have been performed in patients treated with DOAC but with a low thrombotic risk. Studies in those at high thrombotic risk are even rarer.

Our observational study proposes to compare at different times (pre-procedure, intra-procedure and post-procedure admission) the interference of DOACs on the determination of Unfractionated Heparin (UFH) in patients admitted for AF or catheter ALT removal in 25 patients treated with rivaroxaban, 25 patients treated with apixaban, and 25 patients treated with dabigatran, compared to 25 patients treated with VKA.

1. in pre-procedure during the relay by UFH, we will determine the specific anti-Xa activity of UFH independently of AOD by neutralizing in vitro the anti-Xa activity of AOD by filtration.
2. In per-procedure we will determine in these same patients the amount of UFH necessary to obtain a coagulation time measured by the satisfactory activating clotting time (ACT) (≥ 300 sec) to start the procedure. Anti-Xa activity will be performed in parallel to determine whether a correlation can be established between ACT and the specific anti-Xa activity of UFH or residual AOD.
3. We will look for a relationship between the occurrence of hemorrhagic and / or thrombotic events and the concentrations of DOAC and / or UFH in pre- and post-procedure. Patients on VKA with standardized management procedures will be the control group.

This study will determine whether a dose modification of UFH should be considered based on the level of DOAC in the area of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 years and older
* Removal of AF or GAD in the left atrium provided by catheter
* Patient on oral anticoagulant: vitamin K antagonist, apixaban, rivaroxaban or dabigatran
* Patient informed and having given oral consent to participate in the research

Exclusion Criteria:

* Lack of social security affiliation
* Patient under guardianship or with curators
* Patient under state medical aid
* Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients requiring catheter AF/GAD ablation.
  Patients will be recruited during the usual follow-up in cardiology consultation. Patients will be divided into 4 groups depending on the oral anticoagulant used:
  * Vitamin K antagonists (n=25)
  * Apixaban (n=25)
  * Rivaroxaban (n=25)
  * Dabigatran (n=25)
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-07-08 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-12-02 (Actual)

PRIMARY OUTCOMES:
Comparison of the specific anti-Xa activity of UFH (after filtration of the AOD) with the overall anti-Xa activity (without filtration) | 24 months
  Comparison between the 4 groups by a 2-way ANOVA test and evaluation of their relationship by simple regression
Comparison between the 4 groups of UFH bolus doses | 24 months
  Comparison between the 4 groups of UFH bolus doses required to obtain the target ACT by ANOVA or nonparametric assay according to normality of distribution.
The relationship between the specific anti-Xa activity of UFH or DOAC and ACT at different times of the study | 24 months
  The relationship will be evaluated in each group by simple regression and by Bland and Altman graphs.

SECONDARY OUTCOMES:
Correlation between the occurrence of bleeding and/or thrombotic events and pre- and post-procedure DOAC and/or UFH concentrations | 24 months
  Determine whether there is a correlation between the occurrence of bleeding and/or thrombotic events and pre- and post-procedure DOAC and/or UFH concentrations.
Comparison of the specific anti-Xa activity of UFH in groups with and without bleeding complications on the one hand or thrombotic on the other hand | 24 months
  Comparison of the specific anti-Xa activity of UFH in groups with and without bleeding complications on the one hand or thrombotic on the other hand by a Student test or by a nonparametric test (Mann-Whitney) according to the normality of the distribution

CONTACTS AND LOCATIONS:
Overall Officials: Nadine Ajzenberg, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hopital Bichat-Claude Bernard, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided